CLINICAL TRIAL: NCT05832827
Title: First-line Carboplatin/Paclitaxel/Lenvatinib/Pembrolizumab Combination for Previously Untreated Advanced or Recurrent Thymic Carcinomas
Brief Title: First-line CBDCA/PTX/LEN/Pembrolizumab Combination for Previously Untreated Advanced or Recurrent Thymic Carcinomas (Artemis)
Acronym: Artemis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH2109
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Untreated Advanced or Recurrent Thymic Carcinomas
Keywords: thymic carcinoma; pembrolizumab; lenvatinib
MeSH Terms: conditions — Thymoma | interventions — pembrolizumab; lenvatinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MK-3475(Pembrolizumab), Lenvatinib, carboplatin, and paclitaxel (Experimental): Intervention: Carboplatin + paclitaxel + pembrolizumab + lenvatinib for 3 weeks (21 days) as 1 cycle, up to a maximum of 4 cycles in the induction phase. Then, maintenance therapy with pembrolizumab and lenvatinib will be continued until progression or unacceptable adverse events up to 31 cycles.
  Interventions: Drug: MK-3475; Drug: Lenvatinib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: MK-3475 — Pembrolizumab will be administered at a dose of 200 mg by intravenous infusion every 21 days (3 weeks) for up to 35 cycles.
  Other Names: Keytruda/MK-3475 (Pembrolizumab)
Drug: Lenvatinib — Lenvatinib will be administered at a dose of 8 mg orally QD every 21 days (3 weeks) for up to 4 cycles in the induction phase, followed by 20 mg QD for up to 31 cycles in the maintenance phase. Then, further maintenance therapy with lenvatinib will be allowed until progression or unacceptable adverse events.
  Other Names: Lenvima/MK-7902/E7080 (Lenvatinib)
Drug: Carboplatin — Carboplatin will be administered at a dose of AUC 5 intravenously every 21 days (3 weeks) for up to 4 cycles in the induction phase.
  Other Names: CBDCA
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 175 mg/m^2 intravenously every 21 days (3 weeks) for up to 4 cycles in the induction phase.
  Other Names: PTX

SUMMARY:
A phase II, investigator-initiated, non-randomized, open-label, single-arm, multicenter study to evaluate the efficacy and safety of Carboplatin/Paclitaxel/Lenvatinib/Pembrolizumab combination for previously untreated advanced or recurrent thymic carcinomas

DETAILED DESCRIPTION:
This is a phase II, investigator-initiated, non-randomized, open-label, single-arm, multicenter study to evaluate the efficacy and safety of Carboplatin/Paclitaxel/Lenvatinib/Pembrolizumab combination for previously untreated advanced or recurrent thymic carcinomas.

Induction chemotherapy consists of carboplatin + paclitaxel + pembrolizumab + lenvatinib for 3 weeks (21 days) as 1 cycle, up to a maximum of 4 cycles. Then, maintenance therapy with pembrolizumab and lenvatinib will be continued until progression or unacceptable adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older at the time of informed consent, who are pathologically (histologically or cytologically) diagnosed with thymic carcinoma for primary or metastatic thymic lesions, are included. They are preferred to be positive for CD5 or c-KIT by immunohistochemical staining. For those with non-squamous epithelial carcinoma negative for p40 or p63, non-primary cases should be excluded based on their clinical and pathological findings. In addition, those with thymoma are excluded.
2. Patients with unresectable advanced thymic carcinoma (equivalent to stage IVa or IVb of Masaoka-Koga classification), metastatic or recurrent, who have not been treated with systemic cancer chemotherapy.

   Or, in the case of stage III Masaoka-Koga classification, patients who are judged to be incapable of radical resection (R0 resection is not possible due to the combined resection of invasive lesions in surrounding organs (pericardial sac, lung, great vessels, etc.) or who are not eligible for curative treatment with chemoradiotherapy. A history of adjuvant chemotherapy and radiation therapy is acceptable for perioperative adjuvant therapy prior to the finding of recurrence. If platinum-containing cancer chemotherapy has been administered as adjuvant therapy, it is eligible if there is an interval of at least 24 weeks before registration.
3. No symptomatic brain metastases, carcinomatous meningitis, or spinal metastases requiring radiotherapy or surgery
4. No prior history of an antiangiogenetic agent targeting VEGFR for thymic carcinoma
5. Not receiving radiotherapy within 14 days before registration Male participants
6. A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 135 days after the last dose of study treatment and refrain from donating sperm during this period.

   Female participants:
7. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
8. The participant provides written informed consent for the trial
9. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
10. Meet the following criteria for Hepatitis B and C Patients with no history of HBV or HCV infection or who meet the following criteria 10.1 Hepatitis B positive subjects Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have an undetectable HBV viral load prior to registration.

    Participants should remain on anti-viral therapy throughout the study intervention and follow local guidelines for HBV anti-viral therapy post-completion of the study intervention.

    10.2 Participants with a history of HCV infection Participants are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to registration.
11. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin-embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
12. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 14 days before registration.
13. Have adequate organ function as defined in the following table (Table 8). Specimens must be collected within 14 days prior to registration.
14. Have a predicted life expectancy of >12 weeks

Exclusion Criteria:

1. Has diagnosed as thymomas
2. Has related immune-related complications such as myasthenia gravis, pure red cell aplasia, or hypogammaglobulinemia
3. Patients with ECG QT correction interval prolongation or history of such prolongation (patients with QTcF > 480 ms)
4. Has a LVEF below the institutional normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
5. A WOCBP who has a positive urine pregnancy test within 72 hours prior to registration (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
6. Has urine protein ≥1 g/24 hours Note: Participants with proteinuria ≥2+ (≥100 mg/dL) on urine dipstick testing (urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria
7. Has had major surgery within 3 weeks prior to the first dose of study interventions
8. Has clinically significant cardiovascular disease within 12 months from the first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
9. Has any of the following a) to i):

   1. History of interstitial pneumonia or evidence of interstitial lung disease
   2. Uncontrollable autoimmune disease receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy
   3. History or complications of hypertensive crisis or hypertensive encephalopathy
   4. Surgery under general anesthesia within 28 days before registration
   5. History of total gastrectomy
   6. Complication of congenital bleeding predisposition or abnormal coagulation
   7. Complication of Grade 3 or higher gastrointestinal or non-gastrointestinal fistula with CTCAE v5.0
   8. History of Grade 3 or higher bleeding (site not specified) with CTCAE v5.0 within 28 days prior to registration
   9. Blood pressure is not well controlled (with 2 or fewer antihypertensive drugs* 2, systolic blood pressure is 150 mmHg or less and diastolic blood pressure is 90 mmHg or less) *Antihypertensive drugs are counted by the number of compounds
10. Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation.
11. Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
12. Active hemoptysis (bright red blood of at least 0.5 teaspoons) within 3 weeks prior to the first dose of the study drug
13. Has received prior radiotherapy within 14 days before registration. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease
14. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed. Approved COVID-19 vaccines (excluding live vaccines and/or live-attenuated vaccines) are allowed
15. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
16. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug
17. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
18. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening),clinically stable and without the requirement of steroid treatment for at least 14 days prior to the first dose of the study intervention
19. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
20. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with the use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
21. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
22. Has an active infection requiring systemic therapy
23. Has a known history of Human Immunodeficiency Virus (HIV) infection
24. Concurrent active Hepatitis B ( defined as HBsAg positive and detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
27. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. Is expecting to father children within 135 days after the last dose of trial treatment
28. Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) by the Blinded independent review committee | Up to 2 years
  RR is defined as the proportion of patients with the best overall response to complete response (CR) or partial response (PR) as evaluated by the independent review committee according to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  The registration date shall be the starting date, and the period up to the earlier of date determined to be progression or the date of death due to any cause.
Overall Survival Rate (OS) | Up to 2 years
  The period from the registration date to the date of death due to any cause.
Duration of response (DoR) | Up to 2 years
  The progression-free survival rate at 1 year and 2nd year, and median DoR are calculated using the Kaplan-Meier method. The 95% confidence interval for the progression-free survival rate at 1 year and 2nd year is calculated using Greenwood's formula. The 95% confidence interval for the median DoR is determined using the Brookmeyer and Crowley method.
Adverse event rate | Up to 2 years
  In the safety analysis target population, the frequency of the worst grade in all cycles according to the CTCAE v5.0 Japanese translation JCOG version is calculated for each adverse event and discontinuation by adverse events due to protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Okuma, MD, Principal Investigator — National Cancer Center, Japan
Locations (1):
- National Cancer Center Hospital, Chūō, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gandhi L, Garassino MC. Pembrolizumab plus Chemotherapy in Lung Cancer. N Engl J Med. 2018 Sep 13;379(11):e18. doi: 10.1056/NEJMc1808567. No abstract available. PMID 30207917
- [Result] Ferrara N, Gerber HP, LeCouter J. The biology of VEGF and its receptors. Nat Med. 2003 Jun;9(6):669-76. doi: 10.1038/nm0603-669. PMID 12778165
- [Result] Ellis LM, Hicklin DJ. VEGF-targeted therapy: mechanisms of anti-tumour activity. Nat Rev Cancer. 2008 Aug;8(8):579-91. doi: 10.1038/nrc2403. Epub 2008 Jul 3. PMID 18596824
- [Result] Cross MJ, Claesson-Welsh L. FGF and VEGF function in angiogenesis: signalling pathways, biological responses and therapeutic inhibition. Trends Pharmacol Sci. 2001 Apr;22(4):201-7. doi: 10.1016/s0165-6147(00)01676-x. PMID 11282421
- [Result] Lieu C, Heymach J, Overman M, Tran H, Kopetz S. Beyond VEGF: inhibition of the fibroblast growth factor pathway and antiangiogenesis. Clin Cancer Res. 2011 Oct 1;17(19):6130-9. doi: 10.1158/1078-0432.CCR-11-0659. Epub 2011 Sep 27. PMID 21953501
- [Result] Phay JE, Shah MH. Targeting RET receptor tyrosine kinase activation in cancer. Clin Cancer Res. 2010 Dec 15;16(24):5936-41. doi: 10.1158/1078-0432.CCR-09-0786. Epub 2010 Oct 7. PMID 20930041
- [Result] Katsuya Y, Horinouchi H, Asao T, Kitahara S, Goto Y, Kanda S, Fujiwara Y, Nokihara H, Yamamoto N, Watanabe S, Tsuta K, Ohe Y. Expression of programmed death 1 (PD-1) and its ligand (PD-L1) in thymic epithelial tumors: Impact on treatment efficacy and alteration in expression after chemotherapy. Lung Cancer. 2016 Sep;99:4-10. doi: 10.1016/j.lungcan.2016.05.007. Epub 2016 May 12. PMID 27565906
- [Result] Cho J, Kim HS, Ku BM, Choi YL, Cristescu R, Han J, Sun JM, Lee SH, Ahn JS, Park K, Ahn MJ. Pembrolizumab for Patients With Refractory or Relapsed Thymic Epithelial Tumor: An Open-Label Phase II Trial. J Clin Oncol. 2019 Aug 20;37(24):2162-2170. doi: 10.1200/JCO.2017.77.3184. Epub 2018 Jun 15. PMID 29906252
- [Result] Giaccone G, Kim C, Thompson J, McGuire C, Kallakury B, Chahine JJ, Manning M, Mogg R, Blumenschein WM, Tan MT, Subramaniam DS, Liu SV, Kaplan IM, McCutcheon JN. Pembrolizumab in patients with thymic carcinoma: a single-arm, single-centre, phase 2 study. Lancet Oncol. 2018 Mar;19(3):347-355. doi: 10.1016/S1470-2045(18)30062-7. Epub 2018 Jan 26. PMID 29395863
- [Result] Travis WD, Brambilla E, Burke AP, Marx A, Nicholson AG. Introduction to The 2015 World Health Organization Classification of Tumors of the Lung, Pleura, Thymus, and Heart. J Thorac Oncol. 2015 Sep;10(9):1240-1242. doi: 10.1097/JTO.0000000000000663. No abstract available. PMID 26291007
- [Result] Detterbeck FC, Huang J. Overview. J Thorac Oncol. 2011 Jul;6(7 Suppl 3):S1689-90. doi: 10.1097/JTO.0b013e31821e7afe. No abstract available. PMID 21847048
- [Result] Girard N, Lal R, Wakelee H, Riely GJ, Loehrer PJ. Chemotherapy definitions and policies for thymic malignancies. J Thorac Oncol. 2011 Jul;6(7 Suppl 3):S1749-55. doi: 10.1097/JTO.0b013e31821ea5f7. No abstract available. PMID 21847058
- [Result] Detterbeck FC, Stratton K, Giroux D, Asamura H, Crowley J, Falkson C, Filosso PL, Frazier AA, Giaccone G, Huang J, Kim J, Kondo K, Lucchi M, Marino M, Marom EM, Nicholson AG, Okumura M, Ruffini E, Van Schil P; Staging and Prognostic Factors Committee; Members of the Advisory Boards; Participating Institutions of the Thymic Domain. The IASLC/ITMIG Thymic Epithelial Tumors Staging Project: proposal for an evidence-based stage classification system for the forthcoming (8th) edition of the TNM classification of malignant tumors. J Thorac Oncol. 2014 Sep;9(9 Suppl 2):S65-72. doi: 10.1097/JTO.0000000000000290. PMID 25396314
- [Result] Lemma GL, Lee JW, Aisner SC, Langer CJ, Tester WJ, Johnson DH, Loehrer PJ Sr. Phase II study of carboplatin and paclitaxel in advanced thymoma and thymic carcinoma. J Clin Oncol. 2011 May 20;29(15):2060-5. doi: 10.1200/JCO.2010.32.9607. Epub 2011 Apr 18. PMID 21502559
- [Result] Hirai F, Yamanaka T, Taguchi K, Daga H, Ono A, Tanaka K, Kogure Y, Shimizu J, Kimura T, Fukuoka J, Iwamoto Y, Sasaki H, Takeda K, Seto T, Ichinose Y, Nakagawa K, Nakanishi Y; West Japan Oncology Group. A multicenter phase II study of carboplatin and paclitaxel for advanced thymic carcinoma: WJOG4207L. Ann Oncol. 2015 Feb;26(2):363-8. doi: 10.1093/annonc/mdu541. Epub 2014 Nov 17. PMID 25403584
- [Result] Katsuya Y, Fujita Y, Horinouchi H, Ohe Y, Watanabe S, Tsuta K. Immunohistochemical status of PD-L1 in thymoma and thymic carcinoma. Lung Cancer. 2015 May;88(2):154-9. doi: 10.1016/j.lungcan.2015.03.003. Epub 2015 Mar 10. PMID 25799277
- [Result] Katsuya Y, Horinouchi H, Seto T, Umemura S, Hosomi Y, Satouchi M, Nishio M, Kozuki T, Hida T, Sukigara T, Nakamura K, Kuchiba A, Ohe Y. Single-arm, multicentre, phase II trial of nivolumab for unresectable or recurrent thymic carcinoma: PRIMER study. Eur J Cancer. 2019 May;113:78-86. doi: 10.1016/j.ejca.2019.03.012. Epub 2019 Apr 13. PMID 30991261
- [Result] Sato J, Satouchi M, Itoh S, Okuma Y, Niho S, Mizugaki H, Murakami H, Fujisaka Y, Kozuki T, Nakamura K, Nagasaka Y, Kawasaki M, Yamada T, Machida R, Kuchiba A, Ohe Y, Yamamoto N. Lenvatinib in patients with advanced or metastatic thymic carcinoma (REMORA): a multicentre, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):843-850. doi: 10.1016/S1470-2045(20)30162-5. PMID 32502444
- [Result] Girard N, Ruffini E, Marx A, Faivre-Finn C, Peters S; ESMO Guidelines Committee. Thymic epithelial tumours: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v40-55. doi: 10.1093/annonc/mdv277. No abstract available. PMID 26314779
- [Result] Yokoi K, Matsuguma H, Nakahara R, Kondo T, Kamiyama Y, Mori K, Miyazawa N. Multidisciplinary treatment for advanced invasive thymoma with cisplatin, doxorubicin, and methylprednisolone. J Thorac Oncol. 2007 Jan;2(1):73-8. doi: 10.1097/JTO.0b013e31802bafc8. PMID 17410014
- [Result] Nishio M, Horai T, Horiike A, Nokihara H, Yamamoto N, Takahashi T, Murakami H, Yamamoto N, Koizumi F, Nishio K, Yusa W, Koyama N, Tamura T. Phase 1 study of lenvatinib combined with carboplatin and paclitaxel in patients with non-small-cell lung cancer. Br J Cancer. 2013 Aug 6;109(3):538-44. doi: 10.1038/bjc.2013.374. Epub 2013 Jul 16. PMID 23860537
- [Result] Padda SK, Riess JW, Schwartz EJ, Tian L, Kohrt HE, Neal JW, West RB, Wakelee HA. Diffuse high intensity PD-L1 staining in thymic epithelial tumors. J Thorac Oncol. 2015 Mar;10(3):500-8. doi: 10.1097/JTO.0000000000000429. PMID 25402569
- [Result] Giaccone G, Kim C. Durable Response in Patients With Thymic Carcinoma Treated With Pembrolizumab After Prolonged Follow-Up. J Thorac Oncol. 2021 Mar;16(3):483-485. doi: 10.1016/j.jtho.2020.11.003. Epub 2020 Nov 25. PMID 33248322
- [Result] Havel JJ. MEK Inhibitors in Lung Cancer-You Can Teach an Old Drug New Tricks. Cancer Res. 2019 Nov 15;79(22):5699-5701. doi: 10.1158/0008-5472.CAN-19-2590. PMID 31772071
- [Result] Radovich M, Pickering CR, Felau I, Ha G, Zhang H, Jo H, Hoadley KA, Anur P, Zhang J, McLellan M, Bowlby R, Matthew T, Danilova L, Hegde AM, Kim J, Leiserson MDM, Sethi G, Lu C, Ryan M, Su X, Cherniack AD, Robertson G, Akbani R, Spellman P, Weinstein JN, Hayes DN, Raphael B, Lichtenberg T, Leraas K, Zenklusen JC; Cancer Genome Atlas Network; Fujimoto J, Scapulatempo-Neto C, Moreira AL, Hwang D, Huang J, Marino M, Korst R, Giaccone G, Gokmen-Polar Y, Badve S, Rajan A, Strobel P, Girard N, Tsao MS, Marx A, Tsao AS, Loehrer PJ. The Integrated Genomic Landscape of Thymic Epithelial Tumors. Cancer Cell. 2018 Feb 12;33(2):244-258.e10. doi: 10.1016/j.ccell.2018.01.003. PMID 29438696
- [Result] Petrini I, Meltzer PS, Kim IK, Lucchi M, Park KS, Fontanini G, Gao J, Zucali PA, Calabrese F, Favaretto A, Rea F, Rodriguez-Canales J, Walker RL, Pineda M, Zhu YJ, Lau C, Killian KJ, Bilke S, Voeller D, Dakshanamurthy S, Wang Y, Giaccone G. A specific missense mutation in GTF2I occurs at high frequency in thymic epithelial tumors. Nat Genet. 2014 Aug;46(8):844-9. doi: 10.1038/ng.3016. Epub 2014 Jun 29. PMID 24974848
- [Result] Hirai F, Seto T, Inamasu E, Toyokawa G, Yoshida T, Nosaki K, Takenaka T, Yamaguchi M, Takenoyama M, Ichinose Y. Results of S-1-based chemotherapy for platinum (and antrathycline)-refractory advanced thymic carcinoma. Anticancer Res. 2014 Oct;34(10):5743-7. PMID 25275083
- [Result] Shepherd A, Riely G, Detterbeck F, Simone CB 2nd, Ahmad U, Huang J, Korst R, Rajan A, Rimner A. Thymic Carcinoma Management Patterns among International Thymic Malignancy Interest Group (ITMIG) Physicians with Consensus from the Thymic Carcinoma Working Group. J Thorac Oncol. 2017 Apr;12(4):745-751. doi: 10.1016/j.jtho.2016.11.2219. Epub 2016 Nov 19. PMID 27876674
- [Derived] Okuma Y, Nomura S, Sakakibara-Konishi J, Tsukita Y, Murakami S, Hosomi Y, Tambo Y, Kogure Y, Yoshioka H, Tamiya M, Ninomiya K, Iwama E. Artemis: A Multicenter, Open-Label, Single-Arm, Phase II Study to Evaluate the Efficacy and Safety of First-Line Carboplatin/Paclitaxel/Lenvatinib/Pembrolizumab Combination for Previously Untreated Advanced or Recurrent Thymic Carcinomas. Clin Lung Cancer. 2024 Jun;25(4):389-394. doi: 10.1016/j.cllc.2024.02.002. Epub 2024 Feb 8. PMID 38413246